CLINICAL TRIAL: NCT02364232
Title: Effects of Home-based vs. Clinic-based Rehabilitation on Sensorimotor, Cognition, Daily Function, and Participation: Bilateral Training With and Without Mirror Feedback Program
Brief Title: Effects of Home-based vs. Clinic-based Rehabilitation on Sensorimotor, Cognition, Daily Function, and Participation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 103-3962A3
Record Dates: First submitted 2015-01-14; First posted 2015-02-18 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2016-11

CONDITIONS: Chronic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home-based (Experimental): Participants in home-based training graoup will receive 1.5 hours/ day, 3 days a week, for 4 contious weeks at home. Participants will receive 2 training stages, including bilateral training with mirror feedback for 30-45 minutes and functional training for 45-60 minutes. Each training stage hase to include above 2 activities.After the end of the home-based training, a four-week wash-out period followed. Then, patients will receive the clinic-based training for 4 continuous weeks.
  Before and after the treatment, a total of 4 evaluations were conducted, including clinical assessments and blood test (each 9c.c.). One month after the end of the course of treatment will be assessed.
  Interventions: Behavioral: bilateral training with and without mirror feedback
- Clinic-based (Active Comparator): Participants in clinic-based training graoup will receive 1.5 hours/ day, 3 days a week, for 4 contious weeks at home. Participants will receive 2 training stages, including bilateral training with mirror feedback for 30-45 minutes and functional training for 45-60 minutes. Each training stage hase to include above 2 activities.After the end of the clinic-based training, a four-week wash-out period followed. Then, patients will receive the home-based training for 4 continuous weeks.
  Before and after the treatment, a total of 4 evaluations were conducted, including clinical assessments and blood test (each 9c.c.). One month after the end of the course of treatment will be assessed.
  Interventions: Behavioral: bilateral training with and without mirror feedback

INTERVENTIONS:
Behavioral: bilateral training with and without mirror feedback

SUMMARY:
The purpose of this study was to compare the treatment effects of home-based or clinic-based bilateral training with and without mirror feedback programon on physiological markers, sensorimotor, cognition, daily functions, and participation among patients with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* The most recent stroke was between 1 month and 5 years
* No serious cognitive impairment (MMSE≥21)
* FMA score =18-62
* No serious muscle spasticity in shoulder, elbow, wrist and finger (MAS≤3)
* Modified rankin Scale=2 to 4

Exclusion Criteria:

* Aphasia that might interfere with understanding instructions
* Stroke in areas other than the brain and brainstem, such as the cerebellum
* other neurological disease, such as dementia
* Muscle and joint have serious pain and inflammatory swelling in affected side.
* Cannot control hypertension, heart disease and serious throbosis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-09; Primary Completion 2017-04-12 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Fugl-Myer Assessment, FMA | Change from baseline up to 4 weeks immediately after the completion of intervention, and change from 4 weeks up immediately after the completion of intervention up to 3 months after the completion of intervention.
Mini-Mental State Exam, MMSE | Change from baseline up to 4 weeks immediately after the completion of intervention
pinch and grasp dynamometer | Change from baseline up to 4 weeks immediately after the completion of intervention, and change from 4 weeks up immediately after the completion of intervention up to 3 months after the completion of intervention.
Modified Ashworth Scale, MAS | Change from baseline up to 4 weeks immediately after the completion of intervention, and change from 4 weeks up immediately after the completion of intervention up to 3 months after the completion of intervention.
Revised Nottingham Sensory Assessment | Change from baseline up to 4 weeks immediately after the completion of intervention
10-Meter Walking Test, 10MWT | Change from baseline up to 4 weeks immediately after the completion of intervention
Box and Block Test, BBT | Change from baseline up to 4 weeks immediately after the completion of intervention
Wolf Motor Function Test, WMFT | Change from baseline up to 4 weeks immediately after the completion of intervention
Chedoke Arm and Hand Activity Inventory | Change from baseline up to 4 weeks immediately after the completion of intervention
Canadian Occupational Performance Measure, COPM | Change from baseline up to 4 weeks immediately after the completion of intervention
Nottingham Extended Activities of Daily Living, NEADL | Change from baseline up to 4 weeks immediately after the completion of intervention, and change from 4 weeks up immediately after the completion of intervention up to 3 months after the completion of intervention.
ABILHAND Questionnaire | Change from baseline up to 4 weeks immediately after the completion of intervention, and change from 4 weeks up immediately after the completion of intervention up to 3 months after the completion of intervention.
Motor Activity Log, MAL | Change from baseline up to 4 weeks immediately after the completion of intervention, and change from 4 weeks up immediately after the completion of intervention up to 3 months after the completion of intervention.
Actigraphy | Change from baseline up to 4 weeks immediately after the completion of intervention
Stroke Impact Scale, SIS | Change from baseline up to 4 weeks immediately after the completion of intervention, and change from 4 weeks up immediately after the completion of intervention up to 3 months after the completion of intervention.
The World Health Organization Quality of Life -Brief version, WHOQOL-BRE | Change from baseline up to 4 weeks immediately after the completion of intervention
Medical Research Council scale,MRC | Change from baseline up to 4 weeks immediately after the completion of intervention
6 minute walk test | Change from baseline up to 4 weeks immediately after the completion of intervention
The Euroqol Quality of Life Scale | Change from baseline up to 4 weeks immediately after the completion of intervention, and change from 4 weeks up immediately after the completion of intervention up to 3 months after the completion of intervention.
Lawton-Brody IADL Scale | Change from baseline up to 4 weeks immediately after the completion of intervention
Pittsburg Sleep Quality Index | Change from baseline up to 4 weeks immediately after the completion of intervention, and change from 4 weeks up immediately after the completion of intervention up to 3 months after the completion of intervention.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment, MoCA | Change from baseline up to 4 weeks immediately after the completion of intervention
Minnesota Rate of Manipulation Test during dual Task | Change from baseline up to 4 weeks immediately after the completion of intervention
Stroop Test | Change from baseline up to 4 weeks immediately after the completion of intervention
Movement Imagery Questionnaire- Revised, Second Edition, MIQ-RS | Change from baseline up to 4 weeks immediately after the completion of intervention
Kinesthetic and Visual Imagery Questionnaire-10, KVIQ-10 | Change from baseline up to 4 weeks immediately after the completion of intervention
Modified Rankin Scale, mRS | baseline
30 second sit-to-stand test | Change from baseline up to 4 weeks immediately after the completion of intervention
Timed up and go test | Change from baseline up to 4 weeks immediately after the completion of intervention
The stroke self-efficacy questionnaire | Change from baseline up to 4 weeks immediately after the completion of intervention
BDI-II，Beck Depression Inventory II | Change from baseline up to 4 weeks immediately after the completion of intervention

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Chang Gung Memorial Hospital, Kaohsiung County
  - Chang Gung Memorial Hospital, Taoyuan

REFERENCES:
- [Derived] Hsieh YW, Chang KC, Hung JW, Wu CY, Fu MH, Chen CC. Effects of Home-Based Versus Clinic-Based Rehabilitation Combining Mirror Therapy and Task-Specific Training for Patients With Stroke: A Randomized Crossover Trial. Arch Phys Med Rehabil. 2018 Dec;99(12):2399-2407. doi: 10.1016/j.apmr.2018.03.017. Epub 2018 Apr 25. PMID 29702070